CLINICAL TRIAL: NCT03833908
Title: Evaluation of the Performance of MAF-1217 on Surgery Induced DED When Administered Pre-operatively in Patients Undergoing Cataract Surgery
Brief Title: Evaluation of the Performance of MAF-1217 on Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VISUfarma SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VF-OS-002/2018
Record Dates: First submitted 2019-01-31; First posted 2019-02-07 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients receiving MAF-1217 (Experimental): patients receiving MAF-1217 from week -2 to week 2 (preand post-surgery, total 4 weeks), standard antibiotic therapy (ofloxacin) from day -3 before surgery, and standard postoperative treatment (topical steroid, dexamethasone for 10 days + antibiotic, ofloxacin for 7 days) from day 0 (post-surgery.
  Interventions: Device: MAF-1217
- patients receiving just standard antibiotic therapy (No Intervention): patients receiving just standard antibiotic therapy (ofloxacin) from day -3 before surgery, and standard postoperative treatment (topical steroid, dexamethasone for 10 days + antibiotic, ofloxacin 7 days) from day 0 (postsurgery).

INTERVENTIONS:
Device: MAF-1217 — Patients will be enrolled at screening (2 weeks before surgery), then will be randomized with a 1:1 ratio to 2 groups of 23 patients each: A. patients receiving MAF-1217 B. patients receiving just standard antibiotic therapy
  Arms: patients receiving MAF-1217

SUMMARY:
MAF-1217 is meant as the medical device which is to be effective in most forms of DED; therefore, it is expected that study patients benefit from study participation, and can reduce the signs and symptoms of surgery induced DED in patients undergoing cataract surgery, in a TID application pre-surgery.

DETAILED DESCRIPTION:
This is a multicentre, pre-market, open label, randomized, prospective study exploring the performance of MAF-1217 when administered pre-surgery, in reducing the sign and symptoms of post-surgery DED in patients undergoing cataract surgery. Patients will be enrolled 2 weeks before Surgery (screening visit), will undergo cataract surgery (Day 0 - Baseline/Surgery), and then will be seen at week 1 and 2 after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old patients, male and female
2. Patients without diagnosed DED (including subclinical DED) or with mild DED, with BUT >7
3. Normal to mild DED according to OSDI chart
4. Diagnosis of Cataract requiring surgery
5. Wishing to participate in the study and able to sign the ICF
6. Shirmer test > 15 mm /5'
7. No topic ophthalmic medication, including lubricating eyedrops administration for at least 4 days before screening visit.

Exclusion Criteria:

1. Neuropathic causes of dry eye (diabetes, long-standing contact lens wearing, previous ocular herpes infections)
2. Patients with diagnosis of Glaucoma
3. Functional and anatomic eyelid abnormalities,
4. Complicated cataract,
5. Suture affixing during surgery,
6. Use of artificial tears in the month preceding the study visit
7. Coexisting corneal diseases
8. Autoimmune diseases
9. Past or active cicatricial conjunctivitis
10. Past ocular surface burns
11. Keratinization of the eyelid margin
12. Sjogren syndrome
13. History of corneal trauma
14. Pregnant and lactating women
15. Younger than 18 years old patients
16. Inability to self-administer study medications
17. Known allergic sensitivity to any of the devices ingredients, or any other type of allergy
18. Participation in a clinical trial during the 3 months prior to the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
break-up time (BUT) | 1 month
  Difference in the change (with respect to the baseline/surgery visit, V0) in the two arms occurred in break-up time (BUT)

SECONDARY OUTCOMES:
osmolarity | 1 month
  Difference in the change (with respect to the baseline/surgery visit, V0) in the two arms occurred in osmolarity
OSDI score | 1 month
  Difference in the change (with respect to the baseline/surgery visit, V0) in the two arms occurred in OSDI score.
  The OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease.
Schirmer test I | 1 month
  Difference in the change (with respect to the baseline/surgery visit, V0) in the two arms occurred in Schirmer test I (test uses paper strips inserted into the eye for several minutes to measure the production of tears)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università di Firenze, Clinica Oculistica II,, Florence
  - Ospedale San Paolo, ASST Santi Paolo e Carlo, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fogagnolo P, Favuzza E, Marchina D, Cennamo M, Vignapiano R, Quisisana C, Rossetti L, Mencucci R. New Therapeutic Strategy and Innovative Lubricating Ophthalmic Solution in Minimizing Dry Eye Disease Associated with Cataract Surgery: A Randomized, Prospective Study. Adv Ther. 2020 Apr;37(4):1664-1674. doi: 10.1007/s12325-020-01288-z. Epub 2020 Mar 17. PMID 32185729